CLINICAL TRIAL: NCT04348643
Title: Clinical Study of CEA-Targeted CAR-T Therapy in Patients With Relapsed and Refractory CEA+ Cancer
Brief Title: Safety and Efficacy of CEA-Targeted CAR-T Therapy for Relapsed/Refractory CEA+ Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chongqing Precision Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBC017
Record Dates: First submitted 2020-04-14; First posted 2020-04-16 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2022-04

CONDITIONS: Solid Tumor; Lung Cancer; Colorectal Cancer; Liver Cancer; Pancreatic Cancer; Gastric Cancer; Breast Cancer
Keywords: CAR-T; Solid Tumor; Lung Cancer; Colorectal Cancer; Liver Cancer; Pancreatic Cancer; Gastric Cancer; Breast Cancer
MeSH Terms: conditions — Lung Neoplasms; Colorectal Neoplasms; Liver Neoplasms; Pancreatic Neoplasms; Stomach Neoplasms; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CEA+ CAR-T (Experimental): CAR-T cell reinfusion is carried out in 1~3 times
  Interventions: Biological: CEA CAR-T cells

INTERVENTIONS:
Biological: CEA CAR-T cells — CEA-CAR-T cells will be administered intravenously.

SUMMARY:
This is a single arm study to evaluate the efficacy and safety of CEA-targeted CAR-T cells therapy for patients with relapsed/refractory CEA+ Cancer,and obtain the recommended dose and infusion plan.

DETAILED DESCRIPTION:
CEA is a classic tumor marker, especially in more than 80% of colorectal cancer patients. In normal tissue cells, only a small amount of CEA is expressed in the cell membrane of the digestive tract cells, and the CEA is expressed toward the cell cavity under physiological conditions to avoid recognition by CAR-T cells targeting CEA. This is a study to evaluate the efficacy and safety of CEA-targeted CAR-T cells therapy,and obtain the recommended dose and infusion plan.

ELIGIBILITY:
Inclusion Criteria:

1. No gender limitation, age 18-75 years old (including boundary value);
2. Late, metastatic, or recurrent malignant tumors that have received at least first-line standard treatment failure (progressive or intolerable disease, such as surgery, chemotherapy, radiotherapy, targeted therapy, etc.) or lack effective treatment, and the tumor CEA positive expression (tumor CEA positive or serum CEA level> 50ng / ml confirmed by histology or pathology);
3. There are measurable and assessable lesions: the diameter of the lesion under CT or MRI scan is greater than 0.5cm;
4. The expected survival time is more than 12 weeks;
5. KPS≥60 ;
6. No serious mental disorders;
7. The functions of important organs are basically normal:

   1. Blood routine: white blood cells> 2.0 × 10^9 / L, neutrophils> 0.8 × 10^9 / L, lymphocytes> 0.5 × 10^9 / L, platelets> 50 × 10^9 / L, hemoglobin> 90g / L;
   2. Cardiac function: cardiac ultrasound indicates that the cardiac ejection fraction is ≥50%, and there is no obvious abnormality on the electrocardiogram;
   3. Renal function: serum creatinine and urea nitrogen ≤3.0 × ULN;
   4. Liver function: ALT and AST ≤5.0 × ULN; total bilirubin ≤3.0 × ULN;
   5. Blood oxygen saturation> 92%.
8. There are no other serious diseases that conflict with this plan (such as autoimmune diseases, immunodeficiency, organ transplantation);
9. There are no contraindications for apheresis or intravenous blood collection or other cell collection;
10. The patient or his guardian agrees to participate in this clinical trial and sign the ICF, indicating that he understands the purpose and procedures of this clinical trial and is willing to participate in the study.

Exclusion Criteria:

1. Have received CAR-T treatment or other genetically modified cell treatment before screening;
2. Participated in other clinical studies within 1 month before screening;
3. Received the following anti-tumor treatment before screening: received chemotherapy, targeted therapy or other experimental drug treatment within 4 weeks, except for those who have confirmed disease progression after treatment;
4. Have received live attenuated vaccine within 4 weeks before screening;
5. Cerebrovascular accident or seizure occurred within 6 months before signing the ICF;
6. Suffering from any of the following heart diseases:

   1. New York Heart Association (NYHA) stage III or IV congestive heart failure;
   2. Myocardial infarction occurred or received coronary artery bypass graft (CABG) ≤6 months before enrollment;
   3. Clinically significant ventricular arrhythmias, or history of syncope of unknown cause (except for conditions caused by vasovagal or dehydration);
   4. Severe cardiac insufficiency, severe heart valve disease and other cardiovascular system diseases;
7. There are active infections or uncontrollable infections requiring systemic treatment within 2 weeks before screening;
8. Active autoimmune diseases;
9. Suffering from chronic enteritis and / or intestinal obstruction;
10. Suffering from other malignant tumors, in addition to fully treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, local prostate cancer after radical resection, and ductal carcinoma in situ after radical resection;
11. Hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive and peripheral blood hepatitis B virus (HBV) DNA titer detection is greater than the normal range; hepatitis C virus (HCV) antibody positive and peripheral blood hepatitis C Virus (HCV) RNA test is greater than the normal range; human immunodeficiency virus (HIV) antibody positive; syphilis test positive;
12. Women who are pregnant or breastfeeding;
13. The situation that other researchers think is not suitable for participating in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-02-20 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events that related to treatment | 2 years
  Therapy-related adverse events will be recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0)

SECONDARY OUTCOMES:
The response rate of CEA CAR-T treatment in patients with relapse/refractory CEA+ Cancer that treatment by CEA CAR-T cells therapy | 6 months
  The response rate of CEA CAR-T treatment will be recorded and assessed according to the irRECIST Version 1.1
Duration of Response (DOR) of CEA CAR-T treatment in patients with refractory/relapsed CEA+ Cancer | 2 years
  DOR will be assessed from the first assessment of CR/PR/SD to the first assessment of recurrence or progression of the disease or death from any cause
Progress-free survival(PFS) of CEA CAR-T treatment in patients with refractory/relapsed CEA+ Cancer | 2 years
  PFS will be assessed from the first CAR-T cell infusion to death from any cause or the first assessment of progression
Overall survival(OS) of CEA CAR-T treatment in patients with refractory/relapsed CEA+ Cancer | 2 years
  OS will be assessed from the first CAR-T cell infusion to death from any cause
Levels of CEA in Serum | 2 years
  In vivo (Serum) quantity of CEA
Rate of CEA CAR-T cells in peripheral blood | 2 years
  In vivo (peripheral blood) rate of CEA CAR-T cells were determined by means of flow cytometry
Quantity of CEA CAR copies in peripheral blood | 2 years
  In vivo (peripheral blood) quantity of CEA CAR copies were determined by means of qPCR
Levels of IL-6 in Serum | 3 months
  In vivo (Serum) quantity of IL-6
Levels of CRP in Serum | 3 months
  In vivo (Serum) quantity of CRP

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Henan Cancer Hospital, Henan